CLINICAL TRIAL: NCT04305977
Title: Writing to Alleviate Violence Exposure for Transgender Women
Brief Title: Writing to Alleviate Violence Exposure for Transgender Women (WAVE-TW)
Acronym: WAVE-TW
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: There was enrollment in the qualitative phase that proceeded this planned open pilot trial. However, community partner experienced barriers to recruitment and enrollment in the context of COVID and needed prioritize non-research functions.
Sponsor: University of Miami (Other)
Collaborators: Empower U Community Health Center (Unknown); Miami Center for AIDS Research at the University of Miami Miller School of Medicine (Unknown)
Responsible Party: Principal Investigator, Sannisha K Dale, Associate Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20190722
Record Dates: First submitted 2020-03-06; First posted 2020-03-12 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: PTSD; Depression; Virus, Human Immunodeficiency
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WAVE-TW Arm (Other): All participants will receive the WAVE-TW intervention.
  Interventions: Behavioral: WAVE-TW

INTERVENTIONS:
Behavioral: WAVE-TW — The WAVE-TW open pilot trial of the intervention consists of 5 sessions conducted individually with each part participant. Each session lasts approximately 30-50 minutes. The first session will be the LifeSteps Adherence session that focuses on cognitive-behavioral and problem-solving techniques to promote adherence. The next four sessions will be dedicated to trauma writing.

SUMMARY:
WAVE - TW (Writing to Alleviate Violence Exposure for Transgender women living with HIV) is an intervention development study which aims to assess the feasibility and acceptability of a proposed trauma writing and adherence intervention that addresses Post-Traumatic Stress Disorder (PTSD) and depressive symptoms, antiretroviral therapy (ART) adherence and viral suppression among transgender women.

ELIGIBILITY:
Inclusion Criteria:

* Living with HIV
* Age 18 or older
* Detectable viral load within the past year
* Transgender female
* English speaking
* Capable of completing and fully understanding the informed consent process and the study procedures
* History of trauma/abuse

Exclusion Criteria:

* Unable to completely and fully understand the consent process and the study procedures.
* Significant interfering mental health symptoms (e.g., untreated active psychosis, active suicidality with a plan).
* Engaged in an intervention to address trauma symptoms and adherence within the past year

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Percentage of participant satisfaction | Up to 11 months
  Perceptions about the participants' satisfaction with the proposed trauma writing and integrated adherence training intervention. The percentage of participants who report being either satisfied or very satisfied as captured by the Client Satisfaction Survey.
Number of Completed visits | Up to 11 months
  Mean number of visits attended by participants with an attendance rate of 70% or above as an indicator of good attendance.

SECONDARY OUTCOMES:
Change in PTSD symptoms as assessed by the PTSD Checklist for DSM-5 | Baseline, 9 months
  Change in PTSD symptoms will be assessed using the self-reported PTSD Checklist from the Diagnostic and Statistical Manual of Mental Disorders (DSM-5). The questionnaire has 20 items with each item having a scoring range of 0-4 with the higher score indicating increased severity of PTSD symptoms. It has demonstrated good validity/reliability (α = .94). Given the small sample size and the primary aim of the open pilot trial of the intervention, we will cautiously examine the quantitative PTSD symptoms.
Change in Depressive symptoms as assessed by the CES-D Scale | Baseline, 9 months
  Change in depressive symptoms will be assessed using the self-report Center for Epidemiologic Studies Depression (CES-D) Scale. The CES-D is a 20-item measure with a total score ranging from 0-60 with the higher score indicating increased depressive symptoms. Given the small sample size and the primary aim of the open pilot trial of the intervention, we will cautiously examine the quantitative depressive symptoms.
Change in HIV viral load levels | Baseline, Up to 6 months
  Viral suppression will be reported as the change in HIV viral load levels obtained from blood samples.
Number of Participants with Viral load suppression | Up to 6 months
  Viral load suppression will be reported as the number of participants with detectable and not detectable viral load status as confirmed via laboratory testing of blood draw samples.

CONTACTS AND LOCATIONS:
Overall Officials: Sannisha Dale, PhD, Principal Investigator — University of Miami
Locations (1):
- UHealth Don Soffer Clinical Research Building, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No